CLINICAL TRIAL: NCT02761070
Title: A Multicenter Randomized Phase III Study for Recurrent Glioblastoma Comparing Bevacizumab Alone With Dose-dense Temozolomide Followed by Bevacizumab (JCOG1308C, RE-GEND-pIII)
Brief Title: Bevacizumab Alone Versus Dose-dense Temozolomide Followed by Bevacizumab for Recurrent Glioblastoma, Phase III
Acronym: RE-GEND
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyorin University (Other)
Collaborators: Japan Clinical Oncology Group (Other)
Responsible Party: Principal Investigator, Motoo Nagane, Professor, Kyorin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG1308C
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Glioblastoma; Recurrence; Progression
Keywords: glioblastoma; recurrent; dose-dense temozolomide; bevacizumab
MeSH Terms: conditions — Glioblastoma; Recurrence; Disease Progression | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (BEV) alone (Active Comparator): Bevacizumab 10 mg/kg, day 1 div, every 2 weeks
  Interventions: Drug: Bevacizumab
- Dose Dense Temozolomide Followed by BEV (Experimental): Temozolomide (120 mg/m2, po, 7 days on/7 days off, every 2 weeks per cycle) up to 48 cycles. The dose will be escalated to 150 mg/m2 at 3rd cycle if the defined conditions are met throughout the first 2 cycles. At recurrence or progression, bevacizumab alone(10 mg/kg, day 1 div, every 2 weeks)
  Interventions: Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodar; Temodal
  Arms: Dose Dense Temozolomide Followed by BEV
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
The aim of this Phase III study is to evaluate the superiority of dose-dense temozolomide (ddTMZ) followed by bevacizumab at ddTMZ failure for glioblastoma at first recurrence or progression, comparing to bevacizumab alone.

DETAILED DESCRIPTION:
Glioblastoma (GBM), the most frequent malignant primary brain tumor, has yet been incurable despite recent progress on its standard of care using TMZ as the main trunk of initial therapy in the newly diagnosed setting. One of the main reasons accounting for the dismal prognosis would attribute to lack of active therapeutic regimens at recurrence.

Bevacizumab, a humanized monoclonal antibody against cardinal angiogenic factor vascular endothelial growth factor (VEGF), has recently shown efficacy for recurrent GBM, and has been approved in Japan, thereby being a standard care for recurrent GBM. Since there is no effective drugs or regimens developed at bevacizumab failure, insertion of another active drug prior to bevacizumab induction would enhance survival time for patients with recurrent GBM.

In Japan, there are currently only few chemotherapeutic agents approved and available for GBM. Among them rechallenge with alternating dosing of TMZ have shown certain efficacy with acceptable toxicities for patients with TMZ-pretreated recurrent GBM, thus being a good candidate for the regimen used prior to bevacizumab at recurrence.

The present proposal of sequential administration of dose dense TMZ (7/14d) followed by bevacizumab wishes to define a new standard of care for recurrent disease and hopes to identify the subgroups of patients with progressive or recurrent glioblastoma that respond particularly well to dose-dense temozolomide regimens.

This study is carried out as a JCOG Brain Tumor Study Group multicenter randomized phase III trial under approval by Advanced Medical Care B system, Ministry of Health, Labour and Welfare, Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of glioblastoma (including giant cell glioblastoma and gliosarcoma) by WHO2007 criteria.
2. For patients who did not undergo surgery for recurrent disease; pre-registration contrast MRI should confirm; (i)progressive or recurrent glioblastoma; (ii)no evidence of acute or subacute cerebral hemorrhage at enrolment; (iii)presence of a measurable lesion.
3. For patients who underwent surgery for recurrent disease; (i)progressive or recurrent glioblastoma must be confirmed on contrast MRI before reoperation; (ii)glioblastoma or anaplastic astrocytoma must be histologically identified in the tissue resected at reoperation; (iii)presence of measurable lesions is not mandatory on pre-registration contrast MRI (more than 4 days after reoperation); (iv)no MRI evidence of aggravating cerebral hemorrhage.
4. No evidence of tumors in the cerebellum, brain stem, optic nerve, olfactory nerve, and pituitary gland.
5. No evidence of meningeal dissemination or gliomatosis cerebri.
6. Prior treatment for newly-diagnosed glioblastoma (or diffuse astrocytoma (Grade II) or anaplastic astrocytoma (Grade III)) with postoperative TMZ administered concomitantly with radiotherapy (>=54 Gy for <=69 years old; >=30 Gy for >=70 years old) and at least for two cycles (5/28d) as an adjuvant treatment have been given.
7. No history of prior treatment with stereotactic radiotherapy (ex. Gamma-knife/Cyberknife), proton beam irradiation, neutron capture therapy, and chemotherapies except standard dose TMZ and immunotherapy (vaccines, immune checkpoint inhibitors, antibodies etc.), bevacizumab (12 weeks or more after termination of prior upfront bevacizumab use) that were combined with TMZ, and intraoperative placement of carmustine wafers, for glioblastoma (including diffuse astrocytoma (Grade II) and anaplastic astrocytoma (Grade III) at onset) diagnosed with WHO2007 criteria.

   Time periods required from the last day of the prior treatment indicated at registration.

   ①Peptide vaccination, immune checkpoint inhibitors, antibodies: 4 weeks.

   ②Bevacizumab: 12 weeks.
8. More than 90 days after completion of radiotherapy. For those who underwent reoperation, between 21 and 28 days postoperatively.
9. Age between 20 and 75 years at enrolment.
10. Karnofsky Performance Status >= 60 within 14 days before enrolment.
11. No prior treatment with chemotherapy, molecular targeted therapy, or radiotherapy to head and neck area for other malignancies.
12. Adequate organ function.
13. Written informed consent.

Exclusion Criteria:

1. Synchronous or metachronous (within 5 years) malignancy, except for carcinoma in situ or mucosal tumors curatively treated with local therapy
2. Active infection requiring systemic therapy
3. Body temperature >= 38 degrees Celsius at registration
4. Women during pregnancy, possible pregnancy, within 28 days after delivery, or breast-feeding
5. Psychosis or with psychotic symptom
6. Continuous systemic use of immunosuppressant except for steroid
7. Uncontrolled diabetes mellitus
8. Unstable angina within 3 weeks, with a history of myocardial infarction within 6 months, or New York Heart Association (NYHA) class II or greater congestive heart failure
9. Inadequately controlled hypertension (cannot be controlled to a systolic pressure of >= 150 mmHg and a diastolic pressure of >= 100 mmHg)
10. History of symptomatic cerebrovascular disorder (including subarachnoid hemorrhage, cerebral infarction and transient ischemic attack) within 6 months or history of vascular disorder requiring intervention (including venous/arterial thrombosis or embolism and aortic aneurysm) within 6 moths
11. History of grade >= 2 hemoptysis within 28 days
12. History of hemorrhagic tendency (e.g., coagulation disorder) or any grade >= 3 hemorrhage within 28 days
13. History of gastrointestinal perforation, fistula, abdominal abscess or uncontrolled peptic ulcer within 6 months
14. Interstitial pneumonia, pulmonary fibrosis, or severe lung emphysema
15. Severe non-healing wound or traumatic fracture at enrolment
16. Hypersensitivity to Chinese Hamster Ovary-derived drugs or other recombinant antibodies
17. Gadolinium allergy
18. Positive HIV antibody
19. Positive Hepatitis B (HB)s antigen

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-07-11 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Time to event. Up to 2 years from the last patient in.
  Overall survival will be measured from registration until death for any reason. If the patient is alive at last follow-up, the patient will be censored at the last time of confirmation of survival.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time to event. Up to 2 years from the last patient in.
  Progression free will be measured from registration until the first occurrence of progression or death.
6-month progression-free survival (6m-PFS) | 6 months from registration
  Number of patients without progression at 6 months from registration divided by number of all registered
Complete response rate | Through study completion, an average of 1 year
  Complete response rate is defined as the rate of complete response after chemotherapy in cases with measurable lesions through completion/termination of the protocol treatment.
Response rate | Through study completion, an average of 1 year
  Response rate is defined as the rate of complete response/partial response after chemotherapy in cases with measurable lesions through completion/termination of the protocol treatment.
Adverse events | Up to 1 year after completion/termination of the protocol treatment.
  Each adverse event must be graded as the worst grade observed during the entire treatment period of each treatment protocol according to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) up to 1 year.
Serious adverse events | Up to 1 year after completion/termination of the protocol treatment.
  Each serious adverse event must be recorded according to CTCAE v4.0 up to 1 year.
Progression-free survival (PFS) from bevacizumab (BEV) initiation | Time to event from initiation of BEV. Up to 2 years from the last patient in.
  Progression free from BEV initiation will be measured from the day of initiation of BEV until the first occurrence of progression or death.
6-month progression-free survival (6m-PFS) after initiation of bevacizumab (BEV) (Experimental Arm Only) | 6 months from initiation of BEV
  Number of patients without progression at 6 months from the day of initiation of BEV divided by number of all second-line (BEV) treated in Experimental Arm
Overall survival after initiation of bevacizumab (BEV) | Time to event from initiation of BEV. Up to 2 years from the last patient in.
  Overall survival from the day of initiation of BEV until death for any reason. If the patient is alive at last follow-up, the patient will be censored at the last time of confirmation of survival.
MMSE non-deterioration rate | MMSE non-deterioration rates will be calculated at 8 and 24 weeks after initiation of protocol treatment
  The MMSE (Mini Mental Status Examination) non-deterioration rate is calculated from the number of patients who underwent baseline MMSE evaluation prior to initiation of protocol treatment as a denominator and the number of those whose MMSE score (normal (30-24), mild decrease (23-20), intermediate decrease (19-10), severe decrease (9-0)) at 16 weeks improved or maintained from that at baseline as a numerator among all eligible patients.
KPS non-deterioration rate | KPS non-deterioration rates will be calculated at 8 and 24 weeks after initiation of protocol treatment
  The KPS non-deterioration rate is calculated from the number of patients whose KPS was recorded prior to initiation of protocol treatment as a denominator and the number of those whose KPS score at 16 weeks improved or maintained from that at baseline as a numerator among all eligible patients. In case KPS is not recorded, it is considered as deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Motoo Nagane, M.D., Ph.D., Study Chair — Kyorin University Faculty of Medicine, Department of Neurosurgery
Locations (37):
- Japan (37):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Hirosaki University School of Medicine, Hirosaki, Aomori
  - Ehime University Graduate School of Medicine, Shizukawa, Ehime
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University, Morioka, Iwate
  - Tohoku University Graduate School of Medicine, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kansai Medical University, Hirakata, Osaka
  - Osaka University Graduate School of Medicine, Suita, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Dokkyo Medical University, Shimotsuge, Tochigi
  - Tokyo Medical And Dental University, Medical Hospital, Bunkyō-Ku, Tokyo
  - University of Yamanashi, Chuo-shi, Yamanashi
  - Chiba University Hospital, Chiba
  - Kusyu University Graduate School of Medical Sciences, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Kagoshima University Graduate School of Medical and Dental Sciences, Kagoshima
  - Kitasato University School of Medicine, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Graduate School of Medicine, Kyoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
  - Nakamura Memorial Hospital, Sapporo
  - Hokkaido University Graduate School of Medicine, Sapporo
  - Shizuoka Canser Center Hospital, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Nihon University School of Medicine Itabashi Hospital, Tokyo
  - Kyorin University Faculty of Medicine, Department of Neurosurgery, Tokyo
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: No